CLINICAL TRIAL: NCT01450501
Title: Chronic Q-fever in Patients With an Abdominal Aortic Disease (QAAD-study)
Acronym: QAAD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jeroen Bosch Ziekenhuis (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, J.C.J.P. Hagenaars, MD, PhD student, department of Surgery, Jeroen Bosch Ziekenhuis
Other Study IDs: 50-51800-98-013
Record Dates: First submitted 2011-10-06; First posted 2011-10-12 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Q-fever; Aortic Aneurysm, Abdominal; Q Fever; Aneurysm; Vascular Graft Infection
MeSH Terms: conditions — Q Fever; Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue will be investigated using Polymerase Chain Reaction. Serology for C.burnetii will be investigated in blood using Immunofluorecense assay (focus diagnostics).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with vascular chronic Q-fever: All patients with chronic Q-fever and an aneurysm or vascular reconstruction

SUMMARY:
Q-fever is a zoonosis caused by Coxiella burnetii, an intracellular bacterium. Since the epidemic outbreak of acute Q-fever in Holland nearly 4030 people have been registered with the acute form of the disease. Knowing that only 40% of all infected people develop symptoms, the number of infected people (and potential candidates for chronic Q-fever) are much higher. Chronic Q-fever generally manifest itself after a couple of months or years after the primary infection (in 1-5% of all cases). The clinical presentation can be a life-threatening and frequently underdiagnosed disease, as endocarditis, infected aneurysm and vascular prosthesis or chronic Q-fever related to pregnancy and immunecompromised patients. That's why a screening program is started in the endemic area and trace patients with chronic Q-fever. So eventually, a greater group of patients with chronic vascular Q-fever can be described. In addition, there is still no therapeutic guideline for management of chronic Q-fever in patient with a vascular chronic Q-fever.

Patients with an aneurysm or vascular graft will be screened for chronic Q-fever. Patients with chronic Q-fever will be included in a follow-up program, in which additional research and treatment will start. The initial treatment of patients with chronic Q-fever is doxycycline and hydroxychloroquine for at least 18 months. In addition, patients will be monitored in 3-monthly controls, blood samples and imaging will be done. Parameters as complaints, titers, circulating DNA, grow of aneurysm, complications etc. will be investigated.

Ultimately, the current therapeutic guideline for management of C. burnetii will be evaluated if it can also be applied for patients with vascular chronic Q-fever.

DETAILED DESCRIPTION:
Study design:

Prospective observational survey

Domain:

Patients with an abdominal aneurysm or central vascular reconstruction in an endemic area after an outbreak of acute Q-fever.

Data collection:

In Jeroen Bosch Hospital and Bernhoven Hospital all patients with an aneurysm or central vascular reconstruction will be screened for Q-fever. Other hospitals in Holland will only check for Q-fever, if they suspect a patient of having an infected aneurysm or prosthesis.

A patient with chronic Q-fever will enter a multidisciplinary follow-up program. First, a PET/CT-scan will be provided (question; signs of an infected aneurysm/prosthesis)and chronic Q-fever endocarditis will be excluded. The patients will initially be treated with doxycycline 2 dd 100mg and plaquenil 200mg 3dd for at least 18 months. A 3-monthly follow-up will start, in which bloodsample, ultrasounds and PET/CTscan will be performed. Data will be collected in SPSS for analyses.

Definitions; Past resolved Q-fever: Any IgG phase 2 and IgG phase 1 <1:1024 Chronic Q-fever: IgG phase 1 >= 1:1024

ELIGIBILITY:
Inclusion Criteria:

* Patients with an aneurysm of the abdominal aorta or iliac arteries of any size.
* Patients with a central vascular reconstruction, such as EVAR, aortic graft and bifurcation graft.

Exclusion Criteria:

- Patients with a recent central vascular reconstruction (after 1-1-2010) due to a stenoses or occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cohort will be selected from patients with an abdominal aortic disease living in an endemic area after an outbreak of acute Q-fever.
Sampling Method: Probability Sample
Enrollment: 999 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Treatment for patients with vascular chronic Q-fever | 3 years
  The current therapeutic guideline for chronic Q-fever, doxycycline and hydrochloroquine, will now be evaluated in patients with vascular chronic Q-fever

SECONDARY OUTCOMES:
Prevalence past resolved Q-fever | 1 year
Symptomatology in patients with vascular chronic Q-fever | 2 years
Additional value of the PET/CT-scan as diagnostic tool in patients with an infected aneurysm or vascular graft | 1,5 years
Grow of aneurysm in patients with a vascular chronic Q-fever | 3 years
Surgical intervention in patients with vascular chronic Q-fever | 3 years
  What number of patients with C.burnetii vascular infection develop an indication for surgery, why and what sort of prosthesis must be used. If a prosthesis is infected, should it be removed or not.
Mortality | 3 years
Conversion rate to chronic Q-fever | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Julia C.J.P. Hagenaars, MD, Principal Investigator — Jeroen Bosch Hospital
Locations (2):
- Netherlands (2):
  - Jeroen Bosch Hospital, 's-Hertogenbosch, North Brabant
  - Bernhoven Hospital, Veghel/Oss, North Brabant